CLINICAL TRIAL: NCT03997903
Title: IMatinib for PAin in Chronic Treatment of Sickle Cell Anemia (IMPACT SCA): A Pilot Study of Imatinib in Patients With Sickle Cell Anemia and Recurrent Vaso-occlusive Pain
Brief Title: Imatinib for Pain in Sickle Cell Anemia
Acronym: IMPACT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Seethal Jacob, MD, MS, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMPACT SCA
Record Dates: First submitted 2019-06-16; First posted 2019-06-25 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib Intervention (Experimental)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — The starting dose for subjects will be 340 mg/m2/day with a maximum dose of 600 mg daily.
  Patients will receive Imatinib orally once daily for 6 months.

SUMMARY:
In this protocol, the investigators propose to evaluate the biochemical effects of imatinib on sickle red blood cells (RBCs). Patients will be administered imatinib mesylate orally following the guidelines previously established for use of imatinib in other disorders. The biochemical effects of imatinib on sickle RBCs will be examined, including changes in their levels of band 3 tyrosine phosphorylation and the abundances of RBC-derived microparticles in their blood. In addition, the patients will be monitored for symptoms of sickle cell disease (SCD). The investigators expect band 3 tyrosine phosphorylation to decrease dramatically in patients treated with imatinib. The investigators also anticipate a reduction in the numbers of RBC-derived microparticles in circulation (quantitated by assaying the number of glycophorin A positive microparticles in peripheral blood samples by flow cytometry. Most importantly, the investigators expect to see a reduction in the frequency of vaso-occlusive crises, and possibly acute chest syndrome and utilization of opioids. The study duration is planned as 6 months in order to provide adequate time for potential change in the primary endpoints (e.g. percent irreversibly sickled cells).

ELIGIBILITY:
Inclusion Criteria:

1. Age: patients must be ≥18 years of age and ≤25 years of age at the time of study entry.
2. Diagnosis: Patients must have documented diagnosis of sickle cell disease (Hemoglobin SS Disease or S-Beta 0 Thalassemia) by either high pressure liquid chromatography (HPLC) or Hemoglobin Electrophoresis
3. Disease status: Patients must have at least 2 documented episodes of vaso-occlusive pain in the prior year as defined by an acute episode of pain lasting greater than 24 hours, with no medically determined cause other than a vaso-occlusive event that resulted in treatment with oral or parenteral opiates or with a parenteral nonsteroidal anti-inflammatory drug.
4. Performance Level: Karnofsky ≥80 for patients >10 years of age and Lansky ≥80 for patients ≤10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Organ function requirements:

   a. Adequate bone marrow function defined as i. Peripheral absolute neutrophil count (ANC) ≥1000/µL ii. Platelet count ≥100,000/ µL (transfusion independent) b. Adequate renal function defined as i. Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥70 mL/min/1.73 m2 or ii. A serum creatinine based on age/gender c. Adequate Liver Function Defined As: i. Total bilirubin (sum of conjugated + unconjugated) ≤1.5 times upper limit of normal (ULN) for age, and ii. serum glutamate pyruvate transaminase (SGPT or ALT) <2.5 upper limit of normal. For the purpose of this study, the ULN for SGPT is 45 U/L iii. Serum albumin ≥2 g/dL d. Adequate cardiac function defined as: i. Shortening fraction or ejection fraction greater than the institutional norm, and ii. Corrected QT interval ≤450 msec
6. Informed Consent: All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Chronic transfusion protocol.

   a. Patients currently on a chronic transfusion protocol are not eligible
2. Hydroxyurea Intolerance

   a. Patients who are ineligible for hydroxyurea due to persistent marrow suppression (e.g. thrombocytopenia, neutropenia)
3. Pregnancy or Breast-Feeding

   a. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
4. Concomitant Medications

   1. Investigational Drugs: Patients who are currently receiving another investigational drug.
   2. Anti-cancer agents: Patients who are currently receiving other anti-cancer agents.
   3. The following CYP3A4 inducers are prohibited 14 days before the start of imatinib and during the study with imatinib: rifampin, rifabutin, carbamazepine, Phenobarbital, phenytoin, St. John's wort, efavirenz, and tipranavir.
   4. The following CYP3A4 inhibitors are prohibited 7 days before the start of imatinib and during the study with imatinib: azole antifungals (itraconazole, ketoconazole); clarithromycin, erythromycin, diltiazem, verapamil, HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfainavir); delavirdine.
5. Patients who have an uncontrolled infection.
6. Prior use of Imatinib: Patients who have previously received imatinib are not eligible for study.
7. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
8. Patient is < 5 years free of a malignancy. Existence of any other malignant disease is not allowed.
9. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study).
10. Patients with a history of QT prolongation, need for concomitant use of anti-arrhythmics or other agents known to prolong QT interval, or electrolyte derangement that cannot be corrected to within normal limits prior to initiation of study drug.
11. Patients with a family history of sudden cardiac death.
12. Patient has a severe and/or uncontrolled medical disease other than sickle cell disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
13. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
14. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
15. Patient had a major surgery within 2 weeks prior to study entry.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Cincinnati Children's Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 met inclusion criteria. 3 of the participants were on treatment arm and 4 were healthy participants.
Groups:
- Control Group for Blood Draws: Participants who were consented for the purposes of providing blood samples to serve as normal controls for laboratory testing. They did not participate in any other study aspects, nor had data collected related to demographics or laboratory parameters.
Period: Overall Study
Arm/Group | Imatinib Intervention | Control Group for Blood Draws
Started | 3 | 4
Completed | 1 | 4
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected for the Control Group.
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Sickle Cell Genotype: HbSS [Number; unit: participants] | 3
Disease Status [Count of Participants; unit: Participants] — Number of participants with vaso occlusive pain episodes.
  Participants | 3
Performance Level [Count of Participants; unit: Participants] — Number of participants with a Karnofsky performance status greater than or equal to 80.
  The Karnofsky Performance Status is a tool used to assess a patient's functional abilities, particularly in research settings. It ranges from 100 (normal, no complaints) to 0 (death). For this study, we required a baseline Karnofsky score greater than or equal to 80 (normal activity with some symptoms or signs of disease).
  Participants | 3
Organ Function [Count of Participants; unit: Participants] — Number of participants with adequate bone marrow, renal, liver, and cardiac function.
  Participants | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Biochemical Effects - Band 3 Phosphorylation
Description: Percent change in Band 3 Phosphorylation tested in red blood cells. Band 3 is a protein found on the membrane of red blood cells.
Time Frame: Change from baseline Band 3 Phosphorylation at 7 months
Population: Baseline samples for 2 of the 3 participants were processed but were not measurable (possible damage during transportation). 2 of the 3 participants did not have month 7 samples collected. 1 was collected by were not measurable (possible damage during transportation).
Measure: Number
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Amount of Microparticles Released From Red Blood Cells
Description: Change in Microparticles released from red blood cells.
  Microparticles are small vesicles released from red blood cells during aging, stress, or other types of damage that contain various proteins from inside the red blood cell, as well as from its membrane.
Time Frame: change from baseline microparticle release at 7 months
Population: Change in microparticle release from baseline to 7 months was calculated for the one participant that completed the study
Measure: Number; unit: Microparticles per microliter of plasma
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 1
Microparticles per microliter of plasma | -48

3. Primary Outcome: Change in Percent Irreversibly Sickled Cells
Description: Functional RBCs is analyzed by two components, one of which is percent irreversibly sickled cells. The percent of irreversibly sickled cells is measure by ektacytometry.
  Red blood cells that sickle and then cannot revert back to its normal shape are considered irreversibly sickled, increasing the likelihood of adhesion to vessel walls, as well as breakdown or hemolysis. Understanding the point of susceptibility of sickling helps us at what partial pressure of oxygen the red blood cell will sickle. The higher the partial pressure, the more resistant the red blood cell is to sickling/breakdown.
Time Frame: Change from baseline of percent irreversibly sickled cells at 7 months
Population: Only one participant completed 7 months of the study to be analyzed
Measure: Number; unit: percent
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 1
percent | 0.32

4. Primary Outcome: Change in Point of Susceptibility to Sickling by OxygenScan
Description: Functional RBCs is analyzed by two components, one of which is Change in Point of Susceptibility to Sickling. This is measured by OxygenScan.
  The point of susceptibility of sickling shows at what partial pressure of oxygen (mmHg) the red blood cell will sickle. The higher the partial pressure, the more resistant the red blood cell is to sickling/breakdown.
Time Frame: Change from baseline of point of susceptibility of sickling at 7 months
Population: Only 1 participant completed 7 months of the study to be analyzed.
Measure: Number; unit: mmHg
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 1
mmHg | -6.39

5. Secondary Outcome: Number of Instances of Vaso-occlusive Crisis (VOC)
Description: Defined as an acute episode of pain lasting greater than 24 hours, with no medically determined cause other than a vaso-occlusive event that resulted in treatment with oral or parenteral opiate agents and/or parenteral nonsteroidal anti-inflammatory agents. Degree of pain was measured by the standard numerical pain scale (0 being little to no pain, 10 being the worst pain).
Time Frame: Assessed monthly from treatment start up to 7 months
Measure: Number; unit: events
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 3
events | 4

6. Secondary Outcome: Number of Instances of Acute Chest Syndrome (ACS)
Description: Defined as respiratory distress (hypoxia, shortness of breath, chest pain, tachypnea) with evidence of an infiltrate on chest x-ray Measured with clinical evaluation.
Time Frame: Assessed monthly from treatment start up to 7 months
Measure: Number; unit: event
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 3
event | 1

7. Secondary Outcome: Opioid Use
Description: Defined as oral opioid use. Oral use will be documented in pain diary by patient/guardian and reviewed at each visit.
Time Frame: Assessed monthly from treatment start up to 7 months
Population: Data was not analyzed as participants did not utilize the pain diary or were lost-to-follow-up so pain diary data was not obtained.
Measure: Number; unit: units on a scale
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Hospitalizations
Description: Defined as an emergency room or clinic visit resulting in an inpatient admission or observation for a sickle cell-related event (e.g. vaso-occlusive pain, acute chest syndrome, etc).
Time Frame: Assessed monthly from treatment start up to 7 months
Measure: Number; unit: hospitalizations
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 3
hospitalizations | 5

9. Secondary Outcome: Assessment of Toxicities of Imatinib in Patients With Sickle Cell Anemia
Description: Assessment of toxicities based on clinical and laboratory evaluation
Time Frame: Assessed monthly from treatment start up to 7 months
Population: Total number of serious adverse events or adverse events during study participation.
Measure: Number; unit: events
Arm/Group | Imatinib Intervention
Number analyzed (Participants) | 3
events | 21

ADVERSE EVENTS:
Time Frame: 3 years
Description: Systematic Assessment through regular investigator assessment and regular laboratory testing. Adverse events were not collected for the control group as they only provided blood samples to serve as controls during shipment/processing.
Arm/Group | Imatinib Intervention
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Intervention (N=3)
Grade 3 Non Cardiac Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Grade 3 Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Grade 3 Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Intervention (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3)
Nasal Congestion (Ear and labyrinth disorders) | 1 (3)
Alanine Aminotransferase Increased (Hepatobiliary disorders) | 2 (3)
Aspartate Aminotransferase Increased (Hepatobiliary disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (3)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (3)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (3)
Hyperuricemia (Renal and urinary disorders) | 1 (3)
Alkaline Phosphatase Increased (Hepatobiliary disorders) | 1 (3)
Hyperglycemia (Endocrine disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03997903/Prot_SAP_001.pdf